CLINICAL TRIAL: NCT00401700
Title: Acceptability and Feasibility of Influenza Vaccine Administration on the Post-partum Floor Prior to Discharge Home During Flu Season
Brief Title: Influenza Vaccine Postpartum Questionnaire
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 06-190
Record Dates: First submitted 2006-11-17; First posted 2006-11-20 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Influenza; Vaccine; Pregnancy
Keywords: influenza; influenza vaccine; pregnancy
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this trial is to assess the knowledge and attitudes of post-partum women regarding influenza and the use of the influenza vaccine in pregnancy.

DETAILED DESCRIPTION:
Women on our post-partum floor will be approached to complete a questionnaire which will assess their knowledge and attitudes regarding influenza and the use of the influenza vaccine in pregnancy. The study will take place over a 2-month period during influenza season, and at the time when the influenza vaccine becomes available.

ELIGIBILITY:
Inclusion Criteria:

* women admitted to the postpartum floor during the study period

Exclusion Criteria:

* inability to read or understand English

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: pregnant women
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2006-10; Primary Completion 2008-01 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark H Yudin, MD, MSc, Principal Investigator — St. Michael's Hospital (Toronto, Canada)
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada